CLINICAL TRIAL: NCT04202991
Title: An Investigation of the Relationship of Pain With Balance and Gait Impairment in People With Chronic Obstructive Pulmonary Disease
Brief Title: The Relationship Between Pain, Balance and Gait in People With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Teesside University (Other)
Collaborators: South Tees Hospitals NHS Foundation Trust (Other); North Tees and Hartlepool NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Samantha Harrison, Principle Lecturer in Research and Innovation, Teesside University
Other Study IDs: 13418ca
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Balance Impairment; Gait Impairment; Pain
Keywords: COPD, balance, gait, pain
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD with pain: People with COPD who also report pain more often than not over the previous 3 months
  Interventions: Other: Exposure - pain
- COPD with no pain: People with COPD who do not report pain more often than not over the previous 3 months

INTERVENTIONS:
Other: Exposure - pain — Groups are defined by their naturally occurring exposure to pain or not
  Groups: COPD with pain

SUMMARY:
The balance, gait and pain in Chronic Obstructive Pulmonary Disease (COPD) study will aim to investigate the link between balance and gait impairment, and high rates of pain in people with COPD. This cross-sectional observational study will compare balance and gait outcomes for people with COPD who have pain, to those who are pain free.

ELIGIBILITY:
Inclusion Criteria:

* Have a spirometry confirmed diagnosis of COPD as per Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines
* Be 18 years or over at the point of recruitment
* Be able to communicate with good verbal English or use adaptive equipment to communicate.
* Be able to complete test procedures
* Stable COPD (six weeks clear of exacerbation)
* No uncorrected visual or somatosensory disturbance

Exclusion Criteria:

* No other conditions that may affect balance or gait e.g. neurological or vestibular conditions
* Recent exacerbation of COPD (within the last six weeks)
* Unable to provide written informed consent
* Unable to speak English or no translation options available
* Any other acute health conditions that would make activity unsafe e.g. acute infection, unstable cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with COPD referred to, or attending, Pulmonary Rehabilitation at local National Health Service Hospitals/Clinics
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Balance Evaluations Systems Test (BESTest) | 20-30 minutes
  BESTest is a quantitative assessment tool that identifies disordered systems underlying postural control that are responsible for poor functional balance. It was developed for clinicians to differentiate balance problems into six underlying systems that may constrain balance. It was developed from the theoretical understanding of balance control systems based on Bernstein's concept that postural control results from a set of interacting systems. It has 36 items that evaluate performance of 6 balance systems: bio-mechanical constraints, stability limits/verticality, anticipatory responses, postural responses, sensory orientation, and stability in gait. A higher score indicates better balance.

SECONDARY OUTCOMES:
Berg Balance Scale | 5 minutes (for additional items not featured within the BESTest
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. A total score of 56 is available, higher scores indicate better balance.
Gait analysis | 10 minutes
  Temporospatial gait analysis using the 'Gaitrite' walkway.

OTHER OUTCOMES:
30 second sit to stand test | 30 seconds
  The 30 Second Sit to Stand Test is also known as 30 second chair stand test, and tests leg strength and endurance in older adults. A higher number of completed sit to stands in 30 seconds indicates better lower limb endurance.
Peak muscle torque (quadriceps, hamstrings, hip abductors and adductors, ankle plantar flexors and dorsiflexors). | 30 minutes
  Muscle strength testing using the Biodex dynamometer. A higher peak torque in Nm indicates better muscle strength.
PiMax | 5 minutes
  Maximum inspiratory pressure measured by a hand held device that participants take an inward breath in to.
Brief Pain Inventory Short Form | 5 minutes
  The Brief Pain Inventory is a pain questionnaire which measures the severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week. Each item is measured on 0-10 scale, 0 being no pain and 10 being the maximum pain score available.
Physical Activity Scale for the Elderly | 5 minutes
  The Physical Activity Scale for the Elderly (PASE) is a questionnaire that combines information on leisure, household and occupational activity. The PASE assesses the types of activities typically chosen by older adults (walking, recreational activities, exercise, housework, yard work, and caring for others. It uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 to 793, with higher scores indicating greater physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha L Harrison, PhD, Principal Investigator — Teesside University
Locations (2):
- United Kingdom (2):
  - South Tees Hospitals NHS Trust, Middlesbrough
  - North Tees Hospitals NHS Trust, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: Yes
Data will be retained indefinitely in anonymised format and shared on reasonable request
Supporting Information: Study Protocol
Time Frame: Once data has been analysed and available indefinitely
Access Criteria: On request to lead publishing author